CLINICAL TRIAL: NCT03362957
Title: Randomized Placebo-Controlled Single Blinded Study of Geniculate Artery Embolization for Knee Pain Secondary to Osteoarthritis
Brief Title: Geniculate Artery Embolization for Knee Pain Secondary to Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-2701
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Osteo Arthritis Knee
Keywords: embolization; vascular

STUDY DESIGN:
Intervention Model Description: This will be a single-blinded randomized-controlled study of GAE versus placebo in a small population with knee pain secondary to arthritis to determine safety and efficacy. The placebo procedure will be a diagnostic angiogram of the knee, without embolization. Appropriate measures will be taken to ensure patients and nursing staff caring for the patient are blinded to assignment. Each patient will be told at the time of recruitment that they may be randomly assigned to sham, but if after 1 month they have not had symptom improvement, their assigned procedure would be revealed and, if they had undergone a sham procedure, they will be allowed to proceed with embolization.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- GAE Procedure (Experimental): Patients will be randomized to receive the Geniculate Artery Embolization Procedure
  Interventions: Device: Geniculate Artery Embolization
- Sham Procedure (Sham Comparator): Patients will be randomized to a sham procedure.
  Interventions: Diagnostic Test: Sham Procedure
- Crossover Arm (Experimental): If after 1 month patients see no improvement, they will be unblinded and crossover to receive the Geniculate Artery Embolization Procedure
  Interventions: Device: Geniculate Artery Embolization

INTERVENTIONS:
Device: Geniculate Artery Embolization — Gel-Bead Microspheres will be used for geniculate artery embolization (GAE) in subjects with knee osteoarthritis.
  Arms: Crossover Arm; GAE Procedure
Diagnostic Test: Sham Procedure — Patients will receive a sham procedure, which will include a diagnostic angiogram
  Arms: Sham Procedure

SUMMARY:
Purpose: To evaluate embolization as a treatment for OA related knee pain versus placebo to demonstrate the actual effect of embolization on pain and disability.

Participants: There will be 21 subjects enrolled over the age 40 with knee pain secondary to arthritis.

Procedures (methods): This will be a single-blinded randomized-controlled study of GAE versus placebo in a small population with knee pain secondary to arthritis to determine safety and efficacy. Clinical procedures and evaluations will consist of a preoperative screening assessment to determine if the potential study subject meets the inclusion and exclusion criteria, enrollment, surgical procedure for geniculate artery embolization, and follow-up visits at 24 hours, 2 weeks, 1, 3, 6, & 12 months. An MRI may be performed after the 1-month visit.

DETAILED DESCRIPTION:
This will be a single-blinded randomized-controlled study of GAE versus placebo in a small population with knee pain secondary to arthritis to determine safety and efficacy. After Institutional Review Board (IRB) approval of a written informed consent and over, approximately a 24 month duration, N=21 subjects will be recruited. Only subjects ≥ 40 years will be screened for study recruitment. Subjects will be randomized in a 2:1 ratio of GAE:Placebo and will be blinded from study treatment (see flow chart below). The placebo procedure will be a diagnostic angiogram of the knee, without embolization. Appropriate measures will be taken to ensure patients and nursing staff caring for the patient are blinded to assignment. Each patient will be told at the time of recruitment that they may be randomly assigned to sham, but if after 1 month they have not had symptom improvement, their assigned procedure would be revealed and, if they had undergone a sham procedure, they will be allowed to proceed with embolization. This second procedure should be shorter than a complete angiogram and embolization, as the detailed angiogram will not need to be repeated, and therefore both arms will have similar total radiation dose.

Clinical procedures and evaluations will consist of a preoperative screening assessment to determine if the potential study subject meets the inclusion and exclusion criteria, enrollment, surgical procedure for geniculate artery embolization, and follow-up visits at 24 hours, 2 weeks, 1, 3, 6, & 12 months. An MRI may be performed after the 1-month visit.

ELIGIBILITY:
Inclusion Criteria:

Moderate to severe knee pain (visual analog scale (VAS) > 50 mm), and Pain refractory to at least 3 months* of conservative therapies (anti- inflammatory drugs, or physical therapy, or muscle strengthening, or intra- articular injections), and Kellgren-Lawrence grade 1, 2 or 3 on radiograph of the knee.

Exclusion Criteria:

Current local infection, or Life expectancy less than 6 months, or Known advanced atherosclerosis, or Rheumatoid or infectious arthritis, or Prior knee surgery, or Uncorrectable coagulopathy including international normalized ratio (INR) > 2.5 or platelets < 30,000, or Iodine allergy resulting in anaphylaxis, or Renal dysfunction as defined by serum creatinine >1.6 dl/mg or estimated glomerular filtration rate (eGFR) <60 obtained within the past 30 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Isaacson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC Hospitals, Chapel Hill, North Carolina
  - Vascular Institute of Virginia, Woodbridge, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients that received the sham procedure crossed over into the crossover arm.
Groups:
- Sham Procedure First, Then GAE Procedure: Patients will be randomized to a sham procedure.
  Sham Procedure: Patients will receive a sham procedure, which will include a diagnostic angiogram
  If after 1 month patients see no improvement, they will be unblinded and crossover to receive the Geniculate Artery Embolization Procedure
  Geniculate Artery Embolization: Gel-Bead Microspheres will be used for geniculate artery embolization (GAE) in subjects with knee osteoarthritis.
Period: Overall Study
Arm/Group | GAE Procedure | Sham Procedure First, Then GAE Procedure
Started | 14 | 7
Crossover to Receive GAE Procedure | 0 | 7
Completed | 14 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in the sham arm crossed over into the crossover arm so the sham participants and crossover participants are the same baseline characteristics except the VAS and WOMAC where they had new baseline scores following the sham procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | GAE Procedure | Sham Procedure First, Then GAE Procedure | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All participants in the sham arm crossed over into the crossover arm so the sham participants and crossover participants have the same baseline characteristics.
  years | 63.9 (8.4) | 62.9 (7.1) | 63.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All participants in the sham arm crossed over into the crossover arm so the sham participants and crossover participants have the same baseline characteristics.
  Participants
    Female | 12 | 6 | 18
    Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants in the sham arm crossed over into the crossover arm so the sham participants and crossover participants have the same baseline characteristics.
  Participants
    Hispanic or Latino | 2 | 0 | 2
    Not Hispanic or Latino | 11 | 6 | 17
    Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants in the sham arm crossed over into the crossover arm so the sham participants and crossover participants have the same baseline characteristics.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 3 | 5
    White | 11 | 4 | 15
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: All participants in the sham arm crossed over into the crossover arm so the sham participants and crossover participants have the same baseline characteristics.
  Participants
    United States | 14 | 7 | 21
WOMAC [Mean (Standard Deviation); unit: units on a scale] — Western Ontario and McMaster University Osteoarthritis Index (WOMAC) will be used to measure function. This is a score derived from a questionnaire in which the patient answers questions regarding rheumatic symptoms in the subcategories of pain (5 items), stiffness (2 items), and physical function (17 items). Individuals select the level of difficulty they have performing various tasks using a 5 point Likert scale (0=None, 1=Slightly, 3=Very, 4=Extremely). Then, results are scored with a total score (minimum 0; maximum 96). A higher score indicates more difficulty in each of the categories. Population: All patients in the sham arm crossed over to receive the GAE procedure. Their baseline scores following the sham procedure are summarized in a separate row. Participants that had the GAE procedure to start are not crossed over.
  units on a scale
    Baseline for study | 64.9 (16.6) | 70.9 (13.1) | 66.6 (14.4)
    Baseline Following Sham Procedure: number analyzed (Participants) | 0 | 7 | 7
    Baseline Following Sham Procedure |  | 65.9 (11.3) | 65.9 (11.3)
VAS [Mean (Standard Deviation); unit: mm] — The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". Pain will be assessed at each of the patient's follow-up visits and used to measure the change from baseline (prior to the GAE procedure). The investigators will use this to measure if the patient's pain level decreases. Population: All patients in the sham arm crossed over to receive the GAE procedure. Their baseline scores following the sham procedure are summarized in a separate row. Participants that had the GAE procedure to start are not crossed over.
  mm
    Baseline | 13.9 (3.1) | 15.4 (3.5) | 14.3 (3.1)
    baseline following sham procedure: number analyzed (Participants) | 0 | 7 | 7
    baseline following sham procedure |  | 14 (2.7) | 14 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean WOMAC Scores at Month 6
Description: Western Ontario and McMaster University Osteoarthritis Index (WOMAC) will be used to measure function. This is a score derived from a questionnaire in which the patient answers questions regarding rheumatic symptoms in the subcategories of pain (5 items), stiffness (2 items), and physical function (17 items). Individuals select the level of difficulty they have performing various tasks using a 5 point Likert scale (0=None, 1=Slightly, 3=Very, 4=Extremely). Then, results are scored with a total score (minimum 0; maximum 96). A higher score indicates more difficulty in each of the categories.
Time Frame: 6 months following procedure
Population: One participant was excluded from the GAE arm due to increased pain that resulted in additional medication and was excluded from the analysis. All sham participants crossed over to receive treatment after 1 month, thus no 6-month data available for this group. One crossover participant did not have WOMAC data available for the 6 month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 13 | 0 | 6
units on a scale | 29 (25) |  | 26 (31)

2. Primary Outcome: Mean Patient Pain as Measured by VAS at Month 6
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". Pain will be assessed at each of the patient's follow-up visits and used to measure the change from baseline (prior to the GAE procedure). The investigators will use this to measure if the patient's pain level decreases.
Time Frame: 6 months following procedure
Population: One participant was excluded from the GAE arm due to increased pain that resulted in additional medication and was excluded from the analysis. All sham participants crossed over to receive treatment after 1 month, thus no 6-month data available for this group. One patient in the crossover arm did not have VAS data available for the 6 month visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 13 | 0 | 6
mm | 20.3 (25.6) |  | 19.2 (35.3)

3. Secondary Outcome: Number of Participants With Reduction in Medication
Description: Reduction in the number or strength of previously initiated OA medical therapy (e.g. NSAIDs) at 6 months follow-up, which will be summarized using counts.
Time Frame: 12 months following procedure
Population: All participants in the sham arm crossed over 1 month after the sham procedure, thus no 6-month data available for this group.
Measure: Count of Participants; unit: Participants
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 14 | 0 | 7
Participants | 5 | 0 | 1

4. Other Pre Specified Outcome: Number of Patient With Complications
Description: The number and description of complications, adverse events, or poor outcomes (such as no improvement in pain) that are secondary to the GAE procedure, which will be summarized using counts.
Time Frame: 6 months following procedure for the "GAE Procedure" and "Crossover Arm" Arms/Groups and 1 month following procedure for the "Sham Procedure" Arm/Group
Measure: Count of Participants; unit: Participants
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 14 | 7 | 7
Participants | 8 | 2 | 5

5. Primary Outcome: Mean WOMAC Scores at Month 1
Description: as for outcome 1
Time Frame: 1 month following procedure
Population: One participant was excluded from the GAE arm due to increased pain that resulted in additional medication and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 13 | 7 | 7
units on a scale | 34.7 (24) | 65.9 (11.3) | 46.3 (29.6)

6. Primary Outcome: Mean Patient Pain as Measured by VAS at Month 1
Description: as for outcome 2
Time Frame: 1 month following procedure
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 13 | 7 | 7
mm | 30.5 (27.9) | 78.4 (10.2) | 39.8 (31)

7. Primary Outcome: Mean WOMAC Scores at Month 3
Description: as for outcome 1
Time Frame: 3 months following procedure
Population: One participant was excluded from the GAE arm due to increased pain that resulted in additional medication and was excluded from the analysis. One additional participant in this arm did not have data available at the 3 month visit. All sham participants crossed over to receive treatment after 1 month, thus no 3-month data available for this group. One patient in the crossover arm did not have WOMAC data available for the 3 month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 12 | 0 | 6
units on a scale | 19.7 (20.5) |  | 39.5 (27.3)

8. Primary Outcome: Mean Patient Pain as Measured by VAS at Month 3
Description: as for outcome 2
Time Frame: 3 months following procedure
Population: One participant was excluded from the GAE arm due to increased pain that resulted in additional medication and was excluded from the analysis. One additional participant in this arm did not have data available at the 3 month visit. All sham participants crossed over to receive treatment after 1 month, thus no 3-month data available for this group. One patient in the crossover arm did not have VAS data available for the 3 month visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
Number analyzed (Participants) | 12 | 0 | 6
mm | 21.3 (27.9) |  | 41.2 (31.1)

ADVERSE EVENTS:
Time Frame: All adverse events were captured following the Sham procedure for 1 month and for the GAE procedure for the duration of the study, approximately 12 months
Arm/Group | GAE Procedure | Sham Procedure | Crossover Arm
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 8/14 | 2/7 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAE Procedure (N=14) | Sham Procedure (N=7) | Crossover Arm (N=7)
Knee pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 2 (2)
Nausea/Vomiting (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin Ischemia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
bleeding at access site (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03362957/Prot_SAP_000.pdf